CLINICAL TRIAL: NCT00432601
Title: Impact of a Plain Language Prostate Cancer Decision Aid on Decision Making
Brief Title: Testing the Helpfulness of 2 Decision Aids for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 05-283
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: decision aid; prostate cancer; patient-physician communication; decision making; literacy
MeSH Terms: conditions — Prostatic Neoplasms; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients will receive Michigan Cancer Consortium decision aid.
  Interventions: Behavioral: type of decision aid
- Arm 2 (Active Comparator): Patients will receive National Comprehensive Cancer Network decision aid.
  Interventions: Behavioral: type of decision aid

INTERVENTIONS:
Behavioral: type of decision aid — We will be comparing two decision aids (MCC vs. NCCN) in terms of their impact on decision making and patient-physician communication.

SUMMARY:
The purpose of this study is to test different methods for communicating information about prostate cancer treatment to men. The investigators are studying how best to present information so men can make informed decisions about what prostate cancer treatment to undergo.

DETAILED DESCRIPTION:
Background/Rationale: Prostate cancer is the second leading cause of cancer related death among men in the United States, and accounts for 29% of all cancers diagnosed in men. Furthermore, approximately one in six men will be diagnosed with prostate cancer in their lifetime. Thus, 17% of male Veterans will be asked to make a decision about the treatment of their prostate cancer. The burden of this disease is further magnified when one considers that most patients will live for years following their diagnosis and with any adverse effects of therapy. Given that there have been no clinical trials showing that any prostate cancer treatment produces an increased likelihood of survival; men are asked to actively participate in treatment decisions. Previous research has revealed that men are often uninformed about their prostate cancer, particularly African American men and men with lower educational attainment. Thus, it is critical to develop and test decision aids that can help all men (especially men with low literacy skills) make an informed decision.

Objective(s): The goal of the study is to compare the impact of a plain language decision aid (DA) to a conventional DA on prostate cancer patients' decision making experience and communication with their physician.

Methods: This study is a randomized controlled trial. Men undergoing a prostate biopsy will be recruited at the time of biopsy and complete a baseline interview (at pre-biopsy or biopsy appointment). Those patients diagnosed with localized prostate cancer will complete two additional interviews: at physician visit (diagnosis), and 7-10 days following physician visit (phone survey). The treatment discussion between patients and their physician will be audio recorded.

Major characteristics: All men, without a prior history of prostate cancer, undergoing a prostate biopsy will be screened for eligibility and enrolled by the study coordinator. Additional inclusion criteria include ability to speak English, provide informed consent, and have a PSA < 20. Physicians can refuse to allow a patient participate in the study at the time of biopsy. Men will be recruited from 4 VA hospitals (Ann Arbor, Durham, Pittsburgh, and San Francisco) and randomized to receive one of two decision aid booklets (plain language vs. conventional).

Major variables and source(s) of data: All survey data will be collected from either face-to-face or phone interviews. The surveys include measures of literacy, numeracy, anxiety, preference for shared decision making, knowledge, treatment preferences, risk perceptions, perception of patient-physician communication, and confidence and satisfaction with the decision making process. All survey questions were read aloud and responses recorded.

Status: Recruitment began in September 2008 and concluded in May of 2012.

1552 men were approached to participate in the study with 1028 agreeing. 1023 completed the Time 1 interview. Of the 334 subjects eligible to continue with study activities, 285 subjects completed the Time 2 interview (biopsy results visit), and 244 completed the Time 3 phone interview.

ELIGIBILITY:
Inclusion Criteria:

Men undergoing a prostate cancer biopsy at Ann Arbor, Durham, San Francisco, or Pittsburgh VAs. Additional inclusion criteria includes ability to speak English, provide informed consent, and have a PSA < 20.

Exclusion Criteria:

Prior history of prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2008-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fagerlin, PhD MA, Principal Investigator — VA Ann Arbor Healthcare System
Locations (4):
- United States (4):
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Durham, North Carolina
  - Center for Health Equity Research and Promotion, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Levy MH, Back A, Benedetti C, Billings JA, Block S, Boston B, Bruera E, Dy S, Eberle C, Foley KM, Karver SB, Knight SJ, Misra S, Ritchie CS, Spiegel D, Sutton L, Urba S, Von Roenn JH, Weinstein SM. NCCN clinical practice guidelines in oncology: palliative care. J Natl Compr Canc Netw. 2009 Apr;7(4):436-73. doi: 10.6004/jnccn.2009.0031. No abstract available. PMID 19406043

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - MCC: Patients will receive Michigan Cancer Consortium decision aid.
  type of decision aid: We will be comparing two decision aids (MCC vs. NCCN) in terms of their impact on decision making and patient-physician communication.
- Arm 2 - NCCN: Patients will receive National Comprehensive Cancer Network decision aid.
  type of decision aid: We will be comparing two decision aids (MCC vs. NCCN) in terms of their impact on decision making and patient-physician communication.
Period: Time 1 to Time 2
Arm/Group | Arm 1 - MCC | Arm 2 - NCCN
Started | 510 | 512
Completed | 141 (There is large drop-off as only one-third of subjects enrolled were eligible to continue the study) | 144 (There is large drop-off as only one-third of subjects enrolled were eligible to continue the study)
Not Completed | 369 | 368
Period: Time 2 to Time 3
Arm/Group | Arm 1 - MCC | Arm 2 - NCCN
Started | 141 | 144
Completed | 122 | 122
Not Completed | 19 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 510 | 512 | 1022
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.41 (5.86) | 63.14 (6.02) | 63.28 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 510 | 512 | 1022

OUTCOME MEASURES:

1. Primary Outcome: Knowledge
Description: Questions addressed the survival benefit and side effects associated with treatment options for localized prostate cancer.
Time Frame: Results visit (Time 2 - approximately 7-10 days after Time 1)
Measure: Mean (Standard Error); unit: percentage correct on a 12 item scale
Arm/Group | Arm 1 - MCC | Arm 2 - NCCN
Number analyzed (Participants) | 139 | 140
percentage correct on a 12 item scale | 53 (.03) | 48 (.03)

ADVERSE EVENTS:
Description: 1 adverse event occurred prior to randomization to a study arm. A participant fainted while in the process of completing a paper survey. The adverse event was reported to our IRB who determined that it was not related to the research protocol.
Arm/Group | Arm 1 - MCC | Arm 2 - NCCN
Serious Adverse Events (participants affected / at risk) | 0/510 | 0/512
Other Adverse Events (participants affected / at risk) | 1/510 | 0/512
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - MCC (N=510) | Arm 2 - NCCN (N=512)
Seizure (Nervous system disorders) | 1 | 0 — A participant had a seizure while at home completing the Time 3 phone interview.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes